CLINICAL TRIAL: NCT02403037
Title: The Effects of Auricular Acupressure on Chemotherapy-Induced Nausea and Vomiting in Female Breast Cancer Patients: A Pilot Randomized Controlled Trial
Brief Title: Auricular Acupressure for Chemotherapy-Induced Nausea and Vomiting in Female Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Lorna Suen, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20150213001
Record Dates: First submitted 2015-03-19; First posted 2015-03-31 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Breast Neoplasms; Nausea; Vomiting
Keywords: Breast Neoplasms; Auricular Therapy; Acupressure; Chemotherapy; Nausea; Vomiting
MeSH Terms: conditions — Breast Neoplasms; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- True Auricular Acupressure Group (Experimental): Participants in this group will receive standard antiemetics before and during chemotherapy, and a 5-day auricular acupressure treatment protocol for controlling nausea and vomiting during the first cycle of chemotherapy.
  Interventions: Device: True auricular acupressure; Drug: Standard anti-emetic treatment (5-HT3 receptor antagonists and/or Dexamethasone)
- Sham Auricular Acupressure Group (Sham Comparator): Participants in this group will receive standard antiemetic medications before and during chemotherapy, and a 5-day sham auricular acupressure intervention protocol during the first cycle of chemotherapy.
  Interventions: Device: Sham auricular acupressure; Drug: Standard anti-emetic treatment (5-HT3 receptor antagonists and/or Dexamethasone)
- Standard Care Group (Other): Participants in this group will only receive standard anti-emetic treatment before and during chemotherapy.
  Interventions: Drug: Standard anti-emetic treatment (5-HT3 receptor antagonists and/or Dexamethasone)

INTERVENTIONS:
Device: True auricular acupressure — A 5-day auricular acupressure at the specific ear acupoints using vaccaria seeds.
  Other Names: Auricular tape with vaccaria seeds
  Arms: True Auricular Acupressure Group
Device: Sham auricular acupressure — A 5-day sham auricular acupressure at the same acupoints as in the true auricular acupressure arm using Junci Medulla but no pressure will be applied.
  Other Names: Auricular tape with Junci Medulla
  Arms: Sham Auricular Acupressure Group
Drug: Standard anti-emetic treatment (5-HT3 receptor antagonists and/or Dexamethasone) — 5-HT3 receptor antagonists and/or Dexamethasone will be administered to manage chemotherapy-induced nausea and vomiting.
  Other Names: 5-HT3 receptor antagonists and/or Dexamethasone

SUMMARY:
To evaluate the feasibility of a three-parallel-arm, placebo-controlled randomized trial using a standard auricular acupressure protocol for managing nausea and vomiting in a homogenous group of female breast cancer patients undergoing chemotherapy.

The null hypotheses of this study are: (1) There will be no significant difference in acute/delayed nausea and vomiting among groups during the intervention period; (2) There will be no significant difference in anticipatory nausea and vomiting among groups before the second cycle of chemotherapy; (3) There will be no significant difference in quality of life status among groups at the end of the first cycle of chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy-induced nausea and vomiting (CINV) is one of the most common and distressing side-effects among cancer patients undergoing chemotherapy. Despite steady progresses in antiemetic prophylaxis and treatment during the past decades, approximately half of cancer patients receiving moderately to highly emetogenic chemotherapy still experience significant nausea and vomiting. Considering the facts that CINV is difficult to be completely controlled by antiemetics along, healthcare professionals has explored the role of non-pharmacological interventions as adjunctive therapy for controlling CINV. Among which, auricular therapy (AT) is a promising approach but the evidence has still not been concluded.

The aim of this study is to test the feasibility of a randomized controlled trial using auricular acupressure protocol for managing nausea and vomiting in female breast cancer patients undergoing chemotherapy. The objectives of this study will be: (1) to pilot the methodological procedure of the randomized controlled trial using a standard auricular acupressure protocol for controlling CINV; (2) to determine the recruitment rate and attrition rate during the whole study period; (3) to determine the feasibility of the study questionnaires and auricular acupressure protocol to the study participants; (4) to identify potential adverse events associated with auricular acupressure; (5) to preliminarily examine the effects of auricular acupressure on CINV and QoL in female breast cancer patients receiving chemotherapy; (6) to explore patients' experience in completing the trial and receiving the intervention; and (7) to refine the study protocol for a future multicenter, large-scale randomized controlled trial.

A three-parallel-arm, placebo-controlled randomized pilot study will be adopted. One hundred and fourteen breast cancer patients scheduled to receive the first cycle of chemotherapy will be recruited from three provincial hospitals in Fuzhou, China, and will be randomly assigned to one of the three groups: the true AT group, the sham AT group or the standard care group. Participants in the true AT group will receive standard anti-emetic medications plus a 5-day auricular acupressure at the specific ear acupoints, participants in the sham AT group will receive standard anti-emetic medications plus a 5-day auricular acupressure at the same acupoints as in the true AT group without any acupoint stimulation, while participants in the standard care group will only be provided with the standard anti-emetic medications. The feasibility outcomes will be the recruitment rate and consent rate during the recruitment stage, the attrition rate during the whole study period, feasibility of the study questionnaires and auricular acupressure protocol to the study participants, and AT-related adverse events. The future main study outcomes will also be measured including acuteCINV, delayed CINV, anticipatory CINV, and quality of life. After completing the pilot clinical trial, a nested qualitative interview will be conducted to explore participants' experience in completing the trial and receiving the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients aged above 18 years old;
* A diagnosis of breast cancer stage I-III;
* Chemotherapy- naive;
* Auricular therapy-naive;
* Be able to communicate in Chinese mandarin;
* Have at least completed a primary school education;
* Agree to participate in the study and be willing to give written informed consent;
* Be scheduled to receive the first cycle of chemotherapy with moderately-high to highly emetogenic potentials;
* Be provided with standard antiemetic medications during chemotherapy.

Exclusion Criteria:

* Extremely weak, disabled or immunocompromised cancer patients;
* Be unable to follow the study instructions to do AT intervention or other research procedures;
* Have concurrent radiotherapy or other kinds of antineoplastic therapy;
* Currently take part in clinical studies on anti-emetic medications or other kinds of non-pharmacological interventions to control CINV, or other studies which are believed to produce potential interactions with this AT trial;
* Have other health problems which may affect the symptoms of CINV such as gastrointestinal disease, liver disease, migraine, tinnitus and Ménière's disease, etc.;
* Ear skin problems which are not appropriate for auricular acupressure including ear infections, ear scars and rashes, ear frostbite, and ear abscess, etc.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, an average of 1 year and 4 months
  Feasibility outcome
Consent Rate | Through study completion, an average of 1 year and 4 months
  Feasibility outcome
Attrition Rate | Through study completion, an average of 1 year and 4 months
  Feasibility outcome
Feasibility of the Study Questionnaires and Auricular Acupressure Protocol | Through study completion, an average of 1 year and 4 months
  Feasibility outcome
Potential Adverse Events associated with Auricular Acupressure | During the 5-day intervention period
  Feasibility outcome

SECONDARY OUTCOMES:
Occurrence of Acute Vomiting | The 2nd day of the first chemotherapy cycle
  Secondary outcome
Frequency of Acute Vomiting | The 2nd day of the first chemotherapy cycle
  Secondary outcome
Occurrence of Acute Nausea | The 2nd day of the first chemotherapy cycle
  Secondary outcome
Severity of Acute Nausea | The 2nd day of the first chemotherapy cycle
  Secondary outcome
Occurrence of Delayed Vomiting | The 6th day of the first chemotherapy cycle
  Secondary outcome
Frequency of Delayed Vomiting | The 6th day of the first chemotherapy cycle
  Secondary outcome
Occurrence of Delayed Nausea | The 6th day of the first chemotherapy cycle
  Secondary outcome
Severity of Delayed Nausea | The 6th day of the first chemotherapy cycle
  Secondary outcome
Anticipatory Nausea and Vomiting | The 1st day of the second chemotherapy cycle
  The measure is a composite
Quality of Life Status | The 21st day of the first chemotherapy cycle
  Secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Lorna SUEN, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (3):
- China (3):
  - The Second People's Hospital of Fujian Province, Fuzhou, Fujian
  - The First People's Hospital of Fujian Province, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian

REFERENCES:
- [Derived] Tan JY, Molassiotis A, Suen LKP, Liu J, Wang T, Huang HR. Effects of auricular acupressure on chemotherapy-induced nausea and vomiting in breast cancer patients: a preliminary randomized controlled trial. BMC Complement Med Ther. 2022 Mar 24;22(1):87. doi: 10.1186/s12906-022-03543-y. PMID 35331208